CLINICAL TRIAL: NCT05259150
Title: The Health for Hearts United Collaborative
Acronym: HHUC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); University of Georgia (Other)
Responsible Party: Principal Investigator, Penny Ralston, Professor, Dean Emeritus & Director, Center on Better Health, Florida State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00000409
Record Dates: First submitted 2021-11-18; First posted 2022-02-28 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Cardiovascular Disease Risk Reduction
MeSH Terms: interventions — Health

STUDY DESIGN:
Intervention Model Description: effectiveness implementation hybrid Type 3 design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Internal Champion (IC) Strategy (Experimental): In the Planning for Health intervention, the IC implementation strategy will include trainings on transformational leadership principles that address challenges that health leaders face in the church setting to assist them in independently planning the cardiovascular health programming for congregants. Limited assistance from staff will be provided in the Preparing for Health and the Delivery of Health interventions.
  Interventions: Behavioral: Health for Hearts United Planning for Health; Behavioral: Health for Hearts United Preparing for Health; Behavioral: Health for Hearts United Delivery of Health
- Expert Professional (EP) Strategy (Experimental): In the Planning for Health intervention, the EP implementation strategy will include the use of external professionals to assist health leaders in the planning of cardiovascular health programming for congregants. Staff will assist health leaders in the Preparing for Health and the Delivery of Health interventions.
  Interventions: Behavioral: Health for Hearts United Planning for Health; Behavioral: Health for Hearts United Preparing for Health; Behavioral: Health for Hearts United Delivery of Health
- Comparison Group Strategy (Active Comparator): In the Planning for Health intervention, the Comparison Group strategy will include process activities with the health leaders (identification of health leaders, meetings of health leaders, assistance of health leaders with recruitment of congregants for research). Except for data collection, participants (health leaders and congregants) will not be involved in the Preparing for Health or the Delivery of Health interventions.
  Interventions: Other: Health for Hearts United Comparison Group Health Ministry Development

INTERVENTIONS:
Behavioral: Health for Hearts United Planning for Health — Participants (health leaders) receive trainings (three entitled Take Charge of Your Health, Eat Better, & Move Around More) and plan for their health ministry and cardiovascular health program to congregants.
  Arms: Expert Professional (EP) Strategy; Internal Champion (IC) Strategy
Behavioral: Health for Hearts United Preparing for Health — Research participants (church congregants) receive cardiovascular health programming prepared by health leaders that includes the following best practices: Individual Goal Setting, Training, Culturally-tailored Materials, Monitoring Tool & Recognition.
  Arms: Expert Professional (EP) Strategy; Internal Champion (IC) Strategy
Behavioral: Health for Hearts United Delivery of Health — The Organization (church) uses best practices to implement Heart Health activities (annual plans, achievements, plans for the year and practices).
  Arms: Expert Professional (EP) Strategy; Internal Champion (IC) Strategy
Other: Health for Hearts United Comparison Group Health Ministry Development — Participants (health leaders) have meetings to develop the health ministry. Research participants (church congregants) do not receive cardiovascular health program.
  Arms: Comparison Group Strategy

SUMMARY:
This proposed project will determine the effectiveness of Health for Hearts United Collaborative (HHUC) implementation strategies in relation to process outcomes and reducing cardiovascular disease (CVD) risk in African Americans (AAs),examining two possible strategies.

DETAILED DESCRIPTION:
This project will determine the effectiveness of HHUC implementation strategies in relation to process outcomes and reducing CVD risk in AAs, guided by ecological theory, the Consolidated Framework for Implementation Research (CFIR), and the Reach, Effectiveness, Adoption, Implementation and Maintenance (RE-AIM) framework. The HHUC model currently includes three components: governance structure, annual events, and basic support. The investigators propose adding a fourth component that includes one of two possible implementation strategies: 1) an internal champions (IC)-driven strategy that includes two features (leadership development, culturally-tailored planning approaches) or 2) an external change agent (external professionals [EP])-driven strategy without these features. The investigators will pilot and refine the IC and EP-driven implementation strategies using health leaders from four churches in the two-county area by determining feasibility and acceptability. Following the pilot, the investigators will use an effectiveness implementation hybrid Type 3 design to evaluate the IC and EP implementation strategies in relation to process outcomes. The study will be conducted in a two-county area in North Florida, using congregants ((18 years of age and older, n=225) in nine churches: three IC treatment, three EP treatment, and three comparison with delayed comparable activities.

ELIGIBILITY:
Inclusion Criteria:

* African American,
* 18 years of age and older,
* not pregnant in the last six months,
* not hospitalized or having a clinically significant medical condition in the past six months

Exclusion Criteria:

* not being African American,
* under the age of 18,
* pregnant in the last six months,
* hospitalized or having a clinically significant medical condition in the past six months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Participant Reach | 12 months
  Percent of participants that are retained in the intervention which will be computed by dividing the number of participants who complete the intervention by the number who enrolled.
Intervention Adoption | 12 months
  Number of participants who attend intervention sessions which is computed by adding the number of attendees to create total attendance.
Intervention Implementation | 12 months
  Checklist to be developed by the investigators and completed by staff that monitors church health leaders' planning for health ministry development and delivery of program to participants.
Intervention Maintenance | 12 months
  Checklist to be developed by investigators regarding whether or not annual plans are submitted. The instrument will include the list of churches and columns for checking yes or no.

SECONDARY OUTCOMES:
Food choice | 12 months
  Food choice questionnaire which is an 18 item list of foods frequently consumed by African Americans, modified from questionnaires in the literature. Participants respond by indicating if they eat the food item, how frequently (daily, weekly, monthly, yearly, or a few times a year) and serving size (small, medium and large).
Fruit and vegetable intake | 12 months
  National Cancer Institute Fruit and Vegetable Screener is a 10-item instrument that includes respondent assessment of portion size. Scores represent number of servings of fruits and vegetables on a daily basis, ranging from the minimum of zero (0). There is no upper maximum score. The higher the number, the more fruit and vegetable servings consumed daily.
Fat intake | 12 months
  National Cancer Institute Fat Screener is a 16 item instrument that measures percent of energy from fat. Scores can range from 0 percent to 100 percent. The higher percent, the higher percent of energy from fat.
Self-report Physical activity | 12 months
  Yale Physical Activity Scale (YPAS) uses a simple checklist to provide estimates of energy expenditure from activity time (minutes per week) and activity dimensions (e.g., housework, yard work) during a typical day/week. Scores can range from 0 kcal/week minimum to 85,680 kcal/week maximum The higher the kcal/week, the higher the physical activity levels.
Objective physical activity | 12 months
  Wearing of an accelerometer (ActiGraph Corporation, Pensacola, FL) which will be worn on the right hip of each participant for five consecutive days. A wear time of 480 min/day will be used as the criterion for a valid day.
Blood pressure | 12 months
  Three blood pressure readings (systolic and diastolic)
Weight | 12 months
  Weight in kilograms
Height | 12 months
  Height in centimeters
Hip circumference | 12 months
  Measurement of hips in inches using tape measure
Waist circumference | 12 months
  Measurement of waist in inches using tape measure
Abdomen circumference | 12 months
  Measurement of abdomen in inches using tape measure

OTHER OUTCOMES:
Cost of Intervention | 12 months
  Costs associated with implementing intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Center on Better Health and Life for Underserved Populations, Tallahassee, Florida, United States

REFERENCES:
- [Background] Hu FB, Rimm E, Smith-Warner SA, Feskanich D, Stampfer MJ, Ascherio A, Sampson L, Willett WC. Reproducibility and validity of dietary patterns assessed with a food-frequency questionnaire. Am J Clin Nutr. 1999 Feb;69(2):243-9. doi: 10.1093/ajcn/69.2.243. PMID 9989687
- [Background] Willett WC, Sampson L, Stampfer MJ, Rosner B, Bain C, Witschi J, Hennekens CH, Speizer FE. Reproducibility and validity of a semiquantitative food frequency questionnaire. Am J Epidemiol. 1985 Jul;122(1):51-65. doi: 10.1093/oxfordjournals.aje.a114086. PMID 4014201
- See also: Hu FB, Rimm E, Smith-Warner SA, Feskanich D, Stampfer MJ, Ascherio A, Sampson L, Willett WC. Reproducibility and validity of dietary patterns assessed with a food-frequency questionnaire. Am J Clin Nutr. 1999 Feb;69(2):243-9. — https://pubmed.ncbi.nlm.nih.gov/9989687/